CLINICAL TRIAL: NCT03908099
Title: Fit-for-Fertility Multicenter Randomized Controlled Trial: Improving Reproductive, Maternal and Neonatal Outcomes in Obese and Infertile
Brief Title: Fit-for-Fertility Multicenter Randomized Controlled Trial
Acronym: FFF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other); Ferring Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Jean-Patrice Baillargeon, Professor of Medicine, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIHR/PJT-155973
Record Dates: First submitted 2019-04-02; First posted 2019-04-09 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Infertility, Female
Keywords: Lifestyle intervention; Weight loss; Obesity; Infertility; Interdisciplinary program
MeSH Terms: conditions — Obesity; Infertility, Female; Weight Loss; Infertility | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: A pragmatic, multicenter, two-arm, parallel randomized controlled trial comparing the Fit-for-Fertility lifestyle program to usual fertility care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fit-For-Fertility program (Experimental): The experimental intervention will be the Fit-for-Fertility Program alone for the first 6 months, then in combination with usual fertility care for an additional 12 months and thereafter, usual fertility care can continue to be provided alone for a maximum follow-up of 24 months. The lifestyle program is provided for a maximum of 18 months if there is no pregnancy, or otherwise, up to the end of pregnancy or to a total study follow-up of 24 months (whichever comes first).
  Interventions: Behavioral: Fit-For-Fertility program
- Standard of care (Active Comparator): The control intervention will consist of immediate initiation of usual fertility care, as recommended by each fertility specialist, for a maximum of 24 months.
  Interventions: Other: Standard of care

INTERVENTIONS:
Behavioral: Fit-For-Fertility program — The Fit-for-Fertility Program aims at implementing progressive and sustainable lifestyle changes. Participants will attend individual sessions with a dietitian and a kinesiologist every 6 weeks for the first 6 months, then every 8 weeks for the 6 following months, and then every 12 weeks until end of the study. Follow-up by telephone/e-mail will be offered between in-person meetings. These professionals will be trained in motivational counselling skills. Participants will also benefit from weekly group sessions divided into 2 parts: 1) Workshops covering 8 different topics (45 minutes) addressing healthy lifestyle and 2) Supervised classes of physical activity where one of 8 different types of exercise (45 minutes) will be practiced. Women will be required to attend all 8 different sessions within the first 6 months. Pregnant women will be met to set new lifestyle objectives specific to pregnancy, including optimal gestational weight gain based on the Institute of Medicine guidelines.
  Arms: Fit-For-Fertility program
Other: Standard of care — The control intervention will consist of immediate initiation of usual fertility care, as recommended by each fertility specialist, for a maximum of 24 months. The experimental intervention will be the Fit-for-Fertility Program alone for the first 6 months, then in combination with usual fertility care for an additional 12 months and thereafter, usual fertility care can continue to be provided alone for a maximum follow-up of 24 months. The lifestyle program is provided for a maximum of 18 months if there is no pregnancy, or otherwise, up to the end of pregnancy or to a total study follow-up of 24 months (whichever comes first).
  Other Names: Fertilty care
  Arms: Standard of care

SUMMARY:
Infertility affects approximately 10-15% of couples and one of its important modifiable risk factor is obesity, which affects 19% of Canadian women of reproductive age. Accordingly, many organizations have recommended that women should be assisted to adopt a healthy lifestyle prior to conception and maintain it during pregnancy. We therefore propose to conduct a multicenter randomized controlled trial (RCT) assessing the lifestyle intervention Fit-For-Fertility in women with infertility and obesity. Our hypothesis is that the Fit-For-Fertility program is an efficient and low cost solution to improve access to motherhood for women suffering from obesity and infertility.

To test our hypothesis, seven fertility clinics having a good ethnic diversity will participate in this RCT and recruit a total of 408 women with obesity (BMI according to ethnicity) who consult at the fertility clinic. Participants will be randomly allocated to one of these two groups: the intervention group will be invited to participate in the Fit-for Fertility Program alone for 6 months and then in combination with usual fertility treatments; while the control group will receive standard fertility treatments from randomisation. The aim of the Fit-for Fertility Program will be to implement progressive and sustainable lifestyle changes, using 1) individual sessions with a dietitian and a kinesiologist every 6-12 weeks, for a total of 18 months or until the end of pregnancy; and 2) eight educational group sessions. Evaluation visits will take place prior to randomisation and then every 6 months for 18 months. Women who become pregnant will be evaluated early during pregnancy and at 26 weeks of gestation. Clinical outcomes will be assessed after a total follow up of 24 months.

Anticipated contributions: The results of our multicenter RCT will provide important data on the importance of a lifestyle program supporting women with obesity consulting in fertility clinics, in order to improve their fertility and response to ART, as well as helping them to have a healthy baby. This study will also provide valuable information on potential cost savings for individuals and the healthcare system.

DETAILED DESCRIPTION:
1. BACKGROUND

   Infertility affects approximately 10-15% of couples and costs associated with medically assisted reproduction (MAR) are growing, such that equitable access to high quality reproductive care is a challenge for the Canadian health care system. This is especially true for women with obesity. A modifiable risk factor for infertility is obesity (body mass index (BMI) >= 30 kg/m2), which accounts for as many as 19% of Canadian women of reproductive age. Moreover, obesity increases the costs of fertility treatments, reduces their effectiveness and predisposes to several pregnancy and neonatal complications. As important, maternal pre-pregnancy BMI and excessive gestational weight gain were consistently associated with early development of obesity and diabetes in the offspring. Childhood obesity is closely linked to adult obesity, which perpetuates the intergenerational cycle of obesity. Accordingly, we strongly believe that targeting women with obesity prior to conception may be essential to reduce the burden of infertility and MAR costs in Canada, as well as obesity and cardiometabolic diseases.

   To prevent these adverse effects, many organizations have recommended that obese women should be assisted to adopt a healthy lifestyle prior to conception and maintain it during pregnancy. In a recent survey, all women who were obese or overweight and considering pregnancy were interested in adopting a healthy lifestyle pre-conception and 91% reported their willingness to participate in a lifestyle program. However, most Canadian women with obesity do not have access to such targeted lifestyle programs integrated with their fertility care. Our solution is therefore to give these women access to the Fit-for-Fertility Program, an interdisciplinary lifestyle intervention, integrated into the fertility clinic care pathway. This program supports participants in their adoption of sustainable healthy behaviours, prior conception and during pregnancy.

   To fill these gaps, in 2010 Dr. Baillargeon set up the Canadian network on reproductive and maternal health of women with obesity and infertility. Through this network, our team has conducted a CIHR-funded RCT evaluating the impact of the Fit-for-Fertility Program, which was implemented at the fertility clinic of the Centre hospitalier universitaire de Sherbrooke (CHUS), on 130 obese women randomized to 1) Control group: standard fertility treatments right away; or 2) Intervention group: follow the Fit-for-Fertility program alone for 6 months, then in combination with fertility treatments if not pregnant. The analysis of the 108 women who completed at least 6 months in the study (83%) shows that after a maximum follow-up of 18 months and in comparison with the standard fertility treatments (n = 57), the Fit-for-Fertility program (n = 51) significantly increased the rates of total pregnancy (61% vs. 39%, p = 0.02) and spontaneous pregnancy (31% vs. 12%, p = 0.01), as well as a tendency to increase live birth (51% vs. 37%, p = 0.14). Such results from the pilot study are highly clinically significant. The total cost of this intervention was only $870 per participant, as compared to standard fertility care costs averaging $4,400 per woman with obesity in the above-mentioned trial. As such, these preliminary results thus suggest that our low-cost lifestyle intervention for women who are obese and infertile may significantly improve their fertility and reduce the need for expensive MAR. These promising findings provide strong justification for further validation in diverse Canadian populations using a multicenter trial.

   The general goals of our research program are therefore to i) improve the fertility of women with obesity, ii) reduce costs associated with their fertility treatments, and iii) promote the health of mothers and their offspring. To achieve this goal, we ask the question: Does the Fit-for-Fertility Program improve in a cost-effective manner the live birth rate and other fertility outcomes, as well as pregnancy and neonatal outcomes, in women with obesity and infertility who consult a fertility clinic, as compared to usual care?
2. OBJECTIVES

Accordingly, the main objectives of our national multicenter RCT are to:

1. Evaluate the effectiveness of the Fit-for-Fertility Program on fertility and lifestyle outcomes in a diverse Canadian population;
2. Assess costs per live birth and other measures of cost-effectiveness of the program; and
3. Determine the impact of the program on maternal and neonatal health.

3. CENTERS INVOLVED IN THE TRIAL

Six fertility clinics covering Canada from coast to coast and having a good ethnic diversity will participate in this RCT: Olive Fertility Centre in Vancouver, with its Asian population; Omega fertility clinic in Winnipeg, Mount Sinai Hospital in Toronto and Centre hospitalier universitaire (CHU) of Montréal, with large multiethnic communities; and CHU of Sherbrooke and CHU of Québec, smaller centers with mainly Caucasian clientele. All clinics have provided strong support and partnership.

4. RANDOMIZATION

Randomization will occur following the baseline visit (V0), when all eligibility criteria will be available for the candidate. Group allocation will be concealed using on-line computerized randomization with permuted blocks of variable block sizes (2 to 6), stratified by center and PCOS status (yes/no), which decreases fertility and may affect response to the lifestyle intervention. Randomization list will be generated by an independent statistician. Participants will be randomized in two arms using 1:1 ratio. Central randomization will be conducted using a customized web-based program designed for the study. The randomization process will be initiated by the site investigator or delegate who will access the web-based system and enter the patient's confirmation of eligibility and informed consent. The patient's unique study identifier and open-label study treatment allocation will then be electronically delivered to the local site investigator or delegate.

Following randomization, the research staff will inform the fertility care team of their patient's allocation group. If the participant is randomized to the control group, the fertility care team will be informed that their patient can undergo fertility treatments immediately, according to their usual care. On the other hand, if the participant is randomized to the intervention group, the fertility clinic will be notified that the patient will have to postpone any medically assisted reproduction (MAR) procedures for the following 6 months, during which she will be enrolled in the Fit-for-Fertility Program. At the end of this first 6-month period, if the participant is not pregnant, the research staff will contact the fertility clinic team to inform them that the participant can now undergo usual fertility care, in combination with the Fit-for-Fertility Program.

5. FOLLOW-UP

As illustrated in the Study Flow Chart, page ix, research evaluation visits will take place in both groups at baseline and every 6 months for a total of 18 months if no pregnancy occurs. Women who will become pregnant within the first 18 months of follow-up will be evaluated at the beginning of pregnancy and at 24-28 weeks of pregnancy, or up to a total follow-up of 24 months. In our pilot trial, only one participant who became pregnant within 18 months of follow-up delivered after a total follow-up of 24 months. Women who will become pregnant after 18 months of follow-up will not undergo research visits during their pregnancy. All measures and evaluations performed during these research visits are detailed below, in section 8.1, and are listed in the Schedule Table at page x. Patients will be instructed to contact the study team if events occur between visits or phone calls. Importantly, all clinical outcomes will be ascertained with participants and their medical records 24 months after participants' randomization, regardless of the timing of their last research visit and the occurrence of a pregnancy. Pregnancy and neonatal outcomes occurring after 24 months from a pregnancy achieved within 24 months will not be included in the primary analysis of the primary outcome, but will be recorded for secondary analyses.

6. ANALYSES OF THE DATA

6.1 Sample Size

Experts from the Canadian network on reproductive and maternal health of women with obesity and infertility were surveyed, and they concluded that the minimal absolute increase in the 18-month cumulative incidence of live birth (live birth rate) between groups of participants that would change clinical practice must be between 10% and 20%. The only RCT that is similar to our study was published in the NEJM26 and used an increase of 15% for their sample size calculation. Therefore, our initial sample size calculation was based on a 15% absolute difference, an estimated live birth rate of 35% in the control group (from our ongoing RCT), a power of 95% and an alpha level of 5%, and resulted in 293 women per group (nQuery avisor 4.0). Assuming a withdrawal rate of 5% (eligibility criteria violation and loss to follow up), the number of women to recruit was initially defined as 616. In our published protocol, the study power was set at 95% to provide enough power for most of our secondary outcome analyses. However, with the approval of our Steering and Expert Advisory committees, study power for the phase 2 was revised to 85%, which is line with the standard in clinical trials (80-85%). Therefore, our sample size calculation is now based on the same assumptions, but with a 85% power, resulting in 194 women per group. Assuming again a 5% loss to follow-up rate, the total recruitment target is now 408 women. Therefore, each of the 6 clinics will have to recruit 68 participants.

6.2 Statistical Analyses

The main variable of interest will be 24-month live birth cumulative incidence and the primary analyses of interest will be ITT, including all randomized participants with available data and no violation of eligibility criteria. The ITT analyses will be supplemented by per-protocol analyses where women will be excluded if they drop out of the study during the first 6 months. The 24-month cumulative incidences of live birth will be compared between the two arms using the Mantel-Haenszel test with stratification by center and PCOS status. This analysis will be supplemented by a survival analysis (log rank test) where the time to live birth will be used. To assess balance across arms, baseline demographic and clinical data of women will be compared between arms. In the very unlikely event that a substantial imbalance is found, additional analyses will be carried to assess the potential confounding effects of this imbalance, using multiple logistic regression and Cox proportional hazards model.

Similar analyses will be used for other clinical outcome variables, which will be assessed as categories, and continuous variables. Subgroup analyses will be performed based on baseline age, level of obesity, ethnic origins, socio-economic status, the cause of infertility and polycystic ovary syndrome status. A 5% level of significance will be used for all analyses.

7. ANTICIPATED CONTRIBUTIONS

The results of our multicenter RCT will have major scientific impact since they will provide important data on the importance of a lifestyle program supporting women with obesity consulting in fertility clinics, in order to improve their fertility and response to ART as well as helping them to have a healthy baby. This study will also provide valuable information on potential cost savings for individuals and the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

1. Infertility defined as (a) failure to achieve a clinical pregnancy after ≥12 months of regular unprotected sexual intercourse, (b) not conceiving after having tried ≥6 months in women with irregular menstrual cycles or ≥35 years of age; or (c) women with an established cause of infertility;
2. Aged between 18 and 40 years; and
3. Obesity (BMI ≥ 30 kg/m² or 27 kg/m² for Asian and Latin American), or overweight for women with PCOS (BMI ≥ 27 kg/m²).

Exclusion Criteria:

1. Any uncontrolled medical or mental condition that contra-indicates fertility treatments, based on clinical judgment of the fertility specialist;
2. If the only clinically indicated MAR procedure is IVF (e.g. bilateral tubal factor, severe male factor, etc.) or in case of insemination with donor, because natural conception is impossible or highly unlikely;
3. Recurrent spontaneous abortions (>2 miscarriages at less than 22 weeks of gestation) within the last 12 months (with evidence of conception, such as positive β-hCG), because these women do not have difficulty to conceive.
4. Previously diagnosed uncontrolled eating disorder or major depression that would contra-indicate the initiation of a lifestyle intervention;
5. A high level of depressive state, as determined by a score for depression on the Hospital Anxiety and Depression Scale (HADS) ≥ 15, since that would contra-indicate the initiation of a lifestyle intervention;
6. Planning for or past history of bariatric surgery;
7. Planning for or engaging in another intensive lifestyle intervention (that includes face-to-face visits every 8 weeks or less, which would be similar to the intervention tested);
8. Inability to understand the language in which group sessions will be provided in the participating center, i.e. French in Quebec province and English in other provinces; and
9. Planning to be unable to attend research visits at the participating center for the next 18 months, due to moving in another region, for example.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 408 (Estimated)
Dates: Start 2019-04-03 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | 24 months
  Cumulative incidence of live birth, based on medical record/questionnaire.

SECONDARY OUTCOMES:
Fertility Outcomes - Rate of biochemical pregnancy | 24 months
  Confirmed by a positive serum β-hCG), based on medical record.
Fertility Outcomes - Rate of ongoing pregnancy | 24 months
  Viable pregnancy of ≥10 weeks of gestation, based on medical record.
Fertility Outcomes - Rate of spontaneous miscarriage | 24 months
  <22 gestational weeks, based on medical record/questionnaire.
Fertility Outcomes - Rate of multiple gestation | 24 months
  More than one fetal heart beat, based on medical record.
Fertility Outcomes - Rate of spontaneous pregnancy | 24 months
  Without following MAR procedures, based on medical record/questionnaire.
Fertility Outcomes - Rate of pregnancy following MAR procedures | 24 months
  By procedures, based on medical record.
Fertility Outcomes - Doses of fertility medications per participant | 24 months
  required during MAR cycles, based on medical record.
Fertility Outcomes - Number of MAR and/or ART cycles per participant | 24 months
  Number of MAR and/or ART cycles, based on medical record.
Fertility Outcomes - Frequency of embryo transfers | 24 months
  After IVF procedures, based on medical record.
Fertility Outcomes - Frequency of complications due to MAR procedures | 24 months
  All type of complications directly related to MAR, based on medical record.
Lifestyle outcomes - Nutrient intake | 18 months or end of pregnancy
  Using a web-based, food frequency questionnaire.
Lifestyle outcomes - Physical activity behaviours | 18 months or end of pregnancy
  Using the International Physical Activity Questionnaires (IPAQ).
Lifestyle outcomes - Measures of physical activity | 18 months or end of pregnancy
  Daily energy expenditure, time spent in various physical activity intensities and step count, using a blinded Fitbit Flex 2 wristband for 7 consecutive days following the visit.
Lifestyle outcomes - Physical fitness level | 18 months or end of pregnancy
  Using the six-minute walk test.
Lifestyle outcomes - Other lifestyles | 18 months or end of pregnancy
  such as alcohol, tobacco and drugs, using a questionnaire.
Lifestyle outcomes - Sleep duration and quality | 18 months or end of pregnancy
  Using the Pittsburgh Sleep Quality Index.
Lifestyle outcomes - Sleep stages | 18 months or end of pregnancy
  Using the Fitbit Flex 2 wristband.
Lifestyle outcomes - Perceived competence | 18 months or end of pregnancy
  Using the Perceived Competence Scale.
Lifestyle outcomes - Readiness | 18 months or end of pregnancy
  Using a conviction/confidence and readiness questionnaire
Lifestyle outcomes - Anxiety/depression | 18 months or end of pregnancy
  Using the Hospital Anxiety and Depression Scale (HADS).
Anthropometric measures - BMI | 18 months or end of pregnancy
  weight and height will be combined to report BMI in kg/m^2; measures will be performed using a standard calibrated scale and stadiometer.
Anthropometric measures - Fat percentage | 18 months or end of pregnancy
  Using a foot-to-foot bioimpedance scale, in sites having this equipment.
Blood markers - Sex steroids | 18 months or end of pregnancy
  Fasting levels.
Blood markers - Endocrine panel | 18 months or end of pregnancy
  Fasting levels.
Blood markers - Metabolic panel | 18 months or end of pregnancy
  Fasting levels.
Incremental health-related cost-effectiveness ratio of live birth | 24 months
  Using costs questionnaires and other sources of data that will be aggregated at this reported value.
Pregnancy outcomes - Gestational weight gain | 24 months
  estimated by subtracting weight at the research visit closest to the onset of pregnancy from both the weight at the last research visit and the last weight available in the record.
Pregnancy outcomes - Gestational complications | 24 months
  such as gestational diabetes, gestational hypertensive disorders, thromboembolism, preterm birth, late fetal loss, stillbirth and post-partum hospital stay >7 days.
Neonatal outcomes - Birth weight | 24 months
  Based on medical record.
Neonatal outcomes - Apgar score | 24 months
  Based on medical record.
Neonatal outcomes - Hypoglycemia | 24 months
  Based on medical record.
Neonatal outcomes - Jaundice | 24 months
  Based on medical record.
Neonatal outcomes - Birth trauma | 24 months
  Based on medical record.
Neonatal outcomes - Admission to neonatal intensive care unit | 24 months
  Based on medical record.
Neonatal outcomes - Death | 24 months
  Neonatal death up to 28 days of life, based on medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Patrice Baillargeon, MD, MSc, Principal Investigator — Université de Sherbrooke
Locations (5):
- Canada (5):
  - Olive Fertility Centre, Vancouver, British Columbia
  - Mount Sinai Hospital, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Centre hospitalier de l'Université Laval, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belan M, Gelinas M, Carranza-Mamane B, Langlois MF, Morisset AS, Ruchat SM, Lavoie K, Adamo K, Poder T, Gallagher F, Pesant MH, Jean-Denis F, Baillargeon JP; Fit-For-Fertility Study Group. Protocol of the Fit-For-Fertility study: a multicentre randomised controlled trial assessing a lifestyle programme targeting women with obesity and infertility. BMJ Open. 2022 Apr 19;12(4):e061554. doi: 10.1136/bmjopen-2022-061554. PMID 35440463